CLINICAL TRIAL: NCT01180751
Title: 18F-Fluorodeoxyglucose Positron Emission Tomography in Oncology and Neurology
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Manitoba (Other)
Collaborators: Winnipeg Regional Health Authority (Other)
Responsible Party: Dr. Daniel Levin, Winnipeg Regional Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B2010:014
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-07

CONDITIONS: Tumors
Keywords: Positron Emission Tomography; Fluorodeoxyglucose; FDG (18F-Fluorodeoxyglucose); Oncology; Neurology
MeSH Terms: conditions — Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [18F]-Fluorodeoxyglucose (Other): Scanning Procedure: Non-diagnostic Computed Tomography (CT) scan followed by a Diagnostic Positron Emission Tomography (PET) scan.
  Interventions: Radiation: [18F]-Fluorodeoxyglucose

INTERVENTIONS:
Radiation: [18F]-Fluorodeoxyglucose — With each Positron Emission Tomography/Computed Tomography (PET/CT)scan an intravenous administration of radioactive glucose (FDG)is given. This is a weight dependent dosage.
  Other Names: FDG (18F-Fluorodeoxyglucose)

SUMMARY:
This clinical trial is being conducted to study the use of a radioactive glucose tracer as an imaging test [Positron Emission Tomography (PET)scan] in adults who have or are suspected of having cancer and in another group of adults to assess for neurologic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected primary or metastatic tumours
* A neurological presentation consistent with the list of indications
* 18 years of age or older of either sex
* Able to provide written informed consent
* Able to tolerate the physical and logistical requirements of completing a Positron Emission Tomography (PET)scan
* Karnofsky score > 60
* Women who are nursing may be included in the study if they are able to discontinue breast feeding for 12 hours

Exclusion Criteria:

* Age <18 years
* Pregnant women; if there is a possibility of pregnancy, bloodwork will be drawn to definitively establish pregnancy status
* Women who are unwilling or unable to discontinue breast feeding for 12 hours post 18F-Fluorodeoxyglucose(FDG) administration
* Subjects who are medically unstable
* Subjects unwilling to provide informed consent.
* Subjects who exceed the safe weight limit of the Positron Emission Tomography (PET) imaging bed or who cannot fit through the PET scanner bore

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To confirm the diagnostic effectiveness of 18F-Fluorodeoxyglucose(FDG) as compared to the gold standard of histopathological diagnosis. | Three years
  The primary outcomes of sensitivity and accuracy of 18F-Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) studies will be obtained by comparing results of the PET scan with the gold standard of histopathological diagnosis when those results are available. Comparison to correlative imaging follow-up, and assessment of efficacy based on feedback from referring physicians will be used in the absence of pathologic data.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P Levin, BSc,MD,FRCPC, Principal Investigator — Winnipeg Regional Health Authority
Locations (1):
- Great West Life PET/CT Centre, Winnipeg, Manitoba, Canada